CLINICAL TRIAL: NCT07358182
Title: Efficacy and Safety of Trastuzumab-rezetecan in HER2-Positive and HER2-Low Breast Cancer: A Multicenter, Observational, Real-World Study Protocol
Brief Title: Efficacy and Safety of Trastuzumab-rezetecan in HER2-Expressing Breast Cancer
Status: Recruiting | Type: Observational
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Other Study IDs: SYSKY-2025-613-03
Record Dates: First submitted 2026-01-14; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-12

CONDITIONS: Trastuzumab-rezetecan; HER2-low Breast Cancer; HER2-positive Breast Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Trastuzumab-rezetecan Treatment Group
  Interventions: Drug: Trastuzumab-rezetecan Treatment Group

INTERVENTIONS:
Drug: Trastuzumab-rezetecan Treatment Group — Trastuzumab-rezetecan: 4.8 mg/kg (for HER2-positive) or 6.4 mg/kg (for HER2-low) per treatment cycle of 21 days. The dosage is to be adjusted at the discretion of the investigator based on the actual clinical situation.
  All patients will receive treatment with a regimen containing Trastuzumab-rezetecan as determined by the investigator. The regimens for other concomitant medications will be selected by the treating physician based on the patient's individual circumstances.

SUMMARY:
This study is a multicenter, observational, real-world investigation. The research plans to enroll 300 HER2-positive and HER2-low breast cancer patients who meet the inclusion criteria. All patients included in the analysis are currently receiving or are scheduled to receive a treatment regimen containing Trastuzumab-rezetecan. There are no restrictions on the treatment regimen, which is entirely based on the clinician's choice. The study aims to evaluate the efficacy and safety of the treatment regimen containing Trastuzumab-rezetecan.

After completing screening examinations and assessments, eligible patients will enter the study treatment phase. They will receive the treatment regimen containing Trastuzumab-rezetecan and undergo follow-up visits according to the protocol. During the study treatment period, patients will undergo imaging and safety assessments as per clinical routine, with the investigator's assessment serving as the final result. Upon treatment completion or study withdrawal, corresponding safety examinations and imaging assessment data will be collected. For neoadjuvant patients, pathological complete response (pCR) will be assessed post-surgery by pathologists at the participating centers.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years, with pathologically confirmed HER2-positive or HER2-low-expressing breast cancer: HER2-positive is defined as IHC 3+ or IHC 2+ with a positive ISH result; HER2-low-expressing is defined as IHC 1+ or IHC 2+ with a negative ISH result for HER2 amplification; hormone receptor status must be clearly documented.
2. Planned to receive treatment with Trastuzumab-rezetecan for Injection in the neoadjuvant, adjuvant, or advanced/metastatic setting; patients with advanced/metastatic disease must have progressed after at least one prior line of systemic therapy.
3. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-2.
4. Women of childbearing potential must have a negative serum pregnancy test within 28 days prior to enrollment, and both male and female patients must be willing to use a highly effective, medically approved method of contraception during the study and for 1 year after the last dose of the study drug.
5. Non-pregnant and non-lactating female patients.
6. Not concurrently participating in any other ongoing clinical studies. The patient or their legal representative has provided informed consent by signing the informed consent form and is willing and able to comply with scheduled visits, the study treatment plan, laboratory tests, and other trial procedures.

Exclusion Criteria:

1. Any evidence of severe or uncontrolled systemic disease, including uncontrolled hypertension, active bleeding disorders, active infections (such as hepatitis B, hepatitis C, and human immunodeficiency virus), or severely impaired bone marrow reserve or organ function (including hepatic and renal impairment), which, in the investigator's opinion, would significantly alter the risk-benefit balance.
2. At the initiation of treatment with Trastuzumab-rezetecan for Injection, the patient has not recovered from any prior treatment-related toxicity of CTCAE grade >3.
3. Known history of hypersensitivity to Trastuzumab-rezetecan for Injection, its excipients, or drugs with similar chemical structures or classes as Trastuzumab-rezetecan.
4. Patients deemed unsuitable for enrollment by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HER2-positive and HER2-low breast cancer patients, including all those analyzed who are currently receiving or plan to receive a treatment regimen containing Trastuzumab-rezetecan.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2029-06-30 (Estimated); Study Completion 2031-06-30 (Estimated)

PRIMARY OUTCOMES:
Adverse events (AEs) | From the signing of the informed consent form until 30 days after the last dose
  Assessed per NCI-CTCAE v5.0 criteria

SECONDARY OUTCOMES:
Pathological Complete Response(pCR） | Estimated 7 years
  No residual invasive cancer is found upon evaluation of the excised breast tissue and regional lymph nodes
Invasive disease free survival(iDFS) | Estimated 7 years
  Time from randomization to the first occurrence of ipsilateral local/regional invasive recurrence, distant metastasis, contralateral invasive breast cancer, or death from any cause.
Progression-free survival (PFS) | Estimated 7 years
  The date of randomization to the first documented disease progression (per RECIST 1.1) or death due to any cause, whichever occurred first
Objective Response Rate (ORR) | Estimated 7 years
  The percentage of patients with ≥30% tumor shrinkage, as evaluated by investigators per RECIST 1.1 criteria
Clinical Benefit Rate (CBR) | Estimated 7 years
  Sum of complete response [CR], partial response [PR], and SD lasting ≥24 weeks), as assessed by investigators according to RECIST 1.1 criteria
Overall Survival (OS) | Estimated 7 years
  The duration from randomization to death event

CONTACTS AND LOCATIONS:
Locations (1):
- Breast Tumor Center, Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No